CLINICAL TRIAL: NCT03446586
Title: Hereditary Hepatorenal Tyrosinemia Natural History (Multicenter Clinical Study): Registry for Patients With Tyrosinemia Type I in Egypt and the Arab World
Brief Title: Hereditary Hepatorenal Tyrosinemia Natural History in Egypt and the Arab World (Multicenter Clinical Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yassin Abdelghaffar Charity Center for Liver Disease and Research (Other)
Collaborators: Society of Friends of Liver Patients in the Arab World (SLPAW) (Unknown)
Responsible Party: Principal Investigator, Dr. Tawhida Yassin Abdel Ghaffar, Professor, Yassin Abdelghaffar Charity Center for Liver Disease and Research
Other Study IDs: Tyrosinemia Registry E&AW 1
Record Dates: First submitted 2018-02-04; First posted 2018-02-27 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Hereditary Tyrosinemia, Type I
MeSH Terms: conditions — Tyrosinemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Fixed liver block samples & frozen whole blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the registry/repository is to understand the natural history of tyrosinemia in our region and to provide a mechanism to store data and specimens to support the conduct of future research about hereditary tyrosinemia among the Arabs.

DETAILED DESCRIPTION:
The purpose of this study is to create an electronic registry of phenotypic, laboratory information, treatment and outcomes options for tyrosinemia type I. The registry is longitudinal in nature including retrospective clinical data from birth to the most recent encounter with all data entered in chronological fashion. The goals of this registry are the better understanding of the natural history and treatment outcomes of these patients and to determine/evaluate biochemical and clinical parameters for monitoring and prognosis of tyrosinemia type I.

ELIGIBILITY:
Inclusion Criteria:

1. Biochemical or molecular diagnosis of Tyrosinemia Type I.
2. Examined/followed by one of the participating sites.
3. Parental/guardian permission (informed consent) for participation.

Exclusion Criteria:

1. Diagnosis of tyrosinemia has been excluded.
2. Not examined/followed by one of the participating sites.
3. Unwilling to provide informed consent for participation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with tyrosinemia type I seen by one of the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-05 (Estimated); Primary Completion 2023-11-05 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Create a registry for tyrosinemia type I. | 5 Years
  This outcome is a binary 'yes/no' outcome as to whether or not this study can successfully create a repository with the intent to store data and specimens to support the conduct of future research on tyrosinemia type I.

CONTACTS AND LOCATIONS:
Overall Officials: Tawhida Y Abdelghaffar, MD, Principal Investigator — Yassin Abdelghaffar Charity Center for Liver Disease and Research
Locations (1):
- Professor Yassin Abdel Ghaffar Charity Center for Liver Disease and Research, Madīnat an Naşr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No